CLINICAL TRIAL: NCT06646835
Title: The Effect of Stress Ball Application on Anxiety and Fetal Heart Rate in Risk Pregnant Women Before Cesarean Section: A Randomized Controlled Trial
Brief Title: The Effect of Stress Ball Application on Anxiety and Fetal Heart Rate Before Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Nazlı Baltacı, Associate Professor, phD, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: OMU-EYUPOGLU-001
Record Dates: First submitted 2024-10-14; First posted 2024-10-17 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Nursing; Pregnant; Anxiety; Caesarean Section; Fetal Conditions
Keywords: Anxiety; Risky pregnant; Nurse; Stress Ball; Fetal heart rate
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The research will be conducted as a two-group, parallel, randomized, controlled experimental study with a pretest-posttest design.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Pregnant women in the control group will not receive any intervention other than routine general care before cesarean section.
- Intervention Group (Experimental): Pregnant women in the intervention group will be explained how to use the stress ball in the obstetric ward before cesarean section. During the practice, pregnant women will be asked to demonstrate the movements of squeezing and loosening the stress ball to ensure correct use. It will be emphasized to the pregnant women that they should squeeze the ball once after counting to three, inhale when they squeeze the ball, exhale when they loosen their grip and focus only on the ball. In the obstetrics ward, this practice will cover the period starting from the time when the patient is waiting in her room to be taken to the operating room for cesarean section, until she is taken from the preop room to the operating room. In this process, the researcher will monitor whether the stress ball is applied correctly or not. In addition, in order to minimize the risk of infection in the hospital environment, the stress balls used will be disinfected with disposable aseptic wipes before being given
  Interventions: Behavioral: Stress Ball Intervention

INTERVENTIONS:
Behavioral: Stress Ball Intervention — The stress ball is a simple and effective tool for reducing anxiety and relaxation as a non-pharmacological method (Yanes et al., 2018). Due to the limited pharmacological options available for pregnant women to reduce anxiety during cesarean section, alternative, complementary or supportive non-pharmacological methods and low-risk approaches are needed (Baltacı & Başer, 2020). It is thought that squeezing the stress ball may be advantageous in reducing anxiety.
  Arms: Intervention Group

SUMMARY:
This study will be conducted to determine the effect of stress ball application on anxiety and fetal heart rate in risk pregnant women before cesarean section. Women with risk pregnancies randomly assigned to intervention (n=44) and control (n=44) groups in a faculty hospital in Turkey will be included in the study. Pregnant women in the intervention group will be instructed how to use the stress ball in the obstetrics ward before cesarean section. During the practice, pregnant women will be asked to demonstrate the movements of tightening and loosening the stress ball to ensure correct use. It will be emphasized to the pregnant women that they should squeeze the ball once after counting to three, inhale when they squeeze the ball, exhale when they loosen their grip and focus only on the ball. Pregnant women in the control group will not receive any intervention other than routine general care. Data will be collected face-to-face by the researcher based on the self-reports of the pregnant women before cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research,
* Be over 18 years of age,
* Having a medically diagnosed risky condition during pregnancy (diabetes, hypertension, threat of preterm labor, pre-eclampsia, etc.),
* Compliance with at least one of the criteria in the "Ministry of Health Risk Assessment Form for Pregnancy" in the evaluation of current pregnancy,
* Planning a cesarean delivery,
* Being in the last trimester of pregnancy (28 weeks and above)
* Having a single live fetus,
* To be able to read and write Turkish.

Exclusion Criteria:

* A diagnosed psychiatric illness,
* Visual, hearing, speech, physical or mental disability,
* Any communication barriers,
* Cardiovascular disease in the pregnant woman and fetus,
* Fetal distress,
* Fetal anomaly,
* Any physical or medical condition that prevents the use of a stress ball,
* Need for urgent intervention before caesarean section according to the physician.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Woman
Enrollment: 88 (Actual)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
State-Trait anxiety score for anxiety | Anxiety levels will be assessed 5 minutes before intervention and 5 minutes after the end of the intervention.
  The anxiety scale developed by Spielberger et al. in 1970 was designed to measure state and trait anxiety levels of individuals. The Turkish version of this scale was evaluated by Öner and Le Compte in 1983 and its reliability and validity were determined. The scale examines anxiety in two different dimensions: State Anxiety measures the feelings of an individual under a certain moment and condition, while Trait Anxiety refers to the general anxiety level of the individual. Each statement in the scale is a 4-point Likert scale (1-none, 2-somewhat, 3-a lot, 4-completely). Two types of expressions are used in the Spielberger State-Trait Anxiety Scale. Direct expressions indicate negative emotions and inverted expressions indicate positive emotions. Items 1,2,5,8,10,11,15,16,19 and 20 in the Spielberg State Anxiety Scale (SSAS) and items 26,27,30,33,36 and 39 in the Spielberg Trait Anxiety Scale (SSAS) are inverted statements. During the evaluation, after the total weights of the direct
Fetal heart rate | Fetal heart rate levels will be assessed 5 minutes before intervention and 5 minutes after the end of the intervention.
  Fetal heart rate will be measured by fetal hand-held Doppler before and after the intervention.

SECONDARY OUTCOMES:
Pulse rate (beats/minute) | Pulse rate of pregnant women will be assessed 5 minutes before intervention and 5 minutes after the end of the intervention.
  Pulse rate (beats/minute) of pregnant women will be recorded before and after the intervention.
respiration rate (times/minute) | Respiration rate of pregnant women will be assessed 5 minutes before intervention and 5 minutes after the end of the intervention.
  Respiration rate (times/minute) of pregnant women will be recorded before and after the intervention.
systolic and diastolic blood pressure (mmHg) | Systolic and diastolic blood pressure of pregnant women will be assessed 5 minutes before intervention and 5 minutes after the end of the intervention.
  Systolic and diastolic blood pressure (mmHg) of pregnant women will be recorded before and after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Nazlı BALTACI, Assoc. Prof., Study Director — baltacinazli@gmail.com; Elif Eyüpoğlu, Principal Investigator — elifeyupogluu@gmail.com
Locations (1):
- Ondokuz Mayıs University, Samsun, Atakum, Turkey (Türkiye)